CLINICAL TRIAL: NCT01342068
Title: The Effectiveness of Diagnosis and Treatment of Thoracic Outlet Syndrome
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Yasmin Qureshi, MHS, MSPT, Assistant Professor, Nova Southeastern University
Other Study IDs: TOS-Dx and Tx
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-02

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Thoracic outlet syndrome; Osteopathic medicine; Osteopathic Manual Manipulations; OMT; Wright's Test; Adson's Test; Halstead's Maneuver; TOS; Vascular Sonography
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Thoracic Outlet Syndrome (TOS) is a condition causing numbness, tingling and weakness in patient's upper limbs. Symptoms are due to compression and restriction of the nerves and blood vessels (neurovascular bundle) that extend from the neck into the upper limb exerted by a patient's various anatomical structures. Neurovascular bundle compression can result in decreased nerve conduction and blood flow through the arteries supplying structures downstream from the restricted site. These anatomical restrictions include tight scalene muscles in the neck, tightened pectorialis minor muscle in the chest and extra ribs growing from the C7 vertebra.

TOS can be diagnosed by using special tests designed to re-elicit neurovascular bundle compression. Upon obtaining a positive test, the patient can undergo osteopathic manipulative treatments (OMT) to change the anatomical restrictions allowing for a decrease of symptoms and even eradication of the syndrome altogether.

Although diagnosis and treatment of TOS is common in osteopathic medicine, the effectiveness of the diagnostic special tests and treatment has not been thoroughly investigated. This study aims to examine the effectiveness of the special tests (Adson's, Wright's hyperabduction and Halstead maneuver) in diagnosing a change in blood flow through the arteries of the upper arm compared to evaluation with Doppler ultrasound to measure blood flow while the tests are performed. Patients with positive tests will be treated with OMT including myofascial release, soft tissue, and articulation to relieve restricting structures. Upon completion of treatment, the special tests will be performed again along with the Doppler ultrasound to measure blood flow through blood vessels. Results then are analyzed statistically for significance of the ability correctly diagnose and treat TOS symptoms.

Results from this study will contribute towards the validity of teaching special tests in osteopathic medical schools and allow for a non-invasive treatment protocol for patients with TOS.

DETAILED DESCRIPTION:
In today's hectic society it becomes a great disadvantage to individuals when they develop pain and discomfort that decreases their ability to function efficiently. Thoracic Outlet Syndrome (TOS) is a condition that causes pain in the upper extremity, typically extending along the inner aspect of the arm and hand. Other symptoms include weakness, numbness and tingling in the upper extremity. A neurovascular bundle that consists of the brachial plexus, subclavian artery and vein travels from the neck into the arm. TOS symptoms result when the nerves or blood vessels are compressed by the surrounding anatomical structures. In performing this research study, our team would like to improve awareness of TOS to all health care professionals as an entrapment neuropathy and differential diagnosis to neck pain with referred pain. We would also like to bring osteopathic medicine, physical therapy and other paradigms of musculoskeletal manual medicine/therapy together to develop a standardized and valid approach to the diagnosis and treatment of TOS which is not currently available.

There are multiple possible causes of TOS, majority of which results in anatomic restrictions. These possible causes include trauma to the shoulder girdle and more commonly postural disturbances. Individuals with TOS often sit at a computer or desk for an extended period of time for work or school. They develop rounded shoulders and a forward head carriage which changes the length and tone of certain muscles and the relationship of structures in relation to the neurovascular bundle. The anatomic disturbances that contribute and is of the greatest interest to osteopathy includes hypertonicity of the anterior and middle scalene muscles in the neck, hypertonicity of the pectorialis muscle from the upper extremity to the 3-5th ribs, somatic dysfunctions of the clavicle, upper thoracic region and ribs (especially the first rib) (Ward, 2003).

TOS is often the resulting diagnosis after elimination of other possible conditions that cause similar symptoms. These other possible conditions include disc herniations, osteoarthritis, tumors and nerve entrapment syndromes such as carpal tunnel syndrome. Currently discrepancies exist between clinicians about the correct approaches to diagnosis and treatment of TOS. Today's technological advancements can help provide more information about the patient's anatomy, however none can be used for diagnosis alone. MRIs are usually best used for confirmation for the evaluation of the region of interest, however in TOS, findings are frequently inconclusive. One reason for this may be the difficulty to evaluate the extent of a muscle spasm or rib somatic dysfunction and the degree to which it is compressing a nerve structure. (Koknel 2005). X-rays are used to eliminate extra ribs in the cervical region as a cause for symptoms. Anomalous cervical ribs are found in 0.17% to 0.74% each year, however, only 10% of individuals experience TOS symptoms and the onset of these symptoms often relates to cervical spine trauma (Novak, Mackinnon, 2002). The diagnosis of TOS remains to be best based on the patient's subjective complaints, physical examination and the exclusion of other pathologies (Novak, Mackinnon, 2002). Clinical assessment of TOS is best achieved by reproduction of symptoms with compression and special orthopaedic provocative tests that re-produces symptoms based on patient position (Koknel, 2005).

These orthopedic special tests will include:

Wright Test (See picture appendix 2): Wright Test, or Hyperabduction Test, is done by bringing the arm into full abduction with the shoulder externally rotated and the elbow extended while monitoring the radial pulse throughout (Magee DJ, 2008). If there is a decrease or absence of pulse the test is positive showing that axillary artery is compressed by either the pectoralis minor muscle or the coracoid process. (Köknel Talu G, 2005)

Adson Test (See picture appendix 3): For Adson Maneuver the examiner externally rotates and extends the effected arm with the elbow extended while monitoring the radial pulse. The patient is then instructed to rotate the head toward the affected side, extend the neck and take a deep breath and hold it. The absence of disappearance of a pulse indicates a positive test (Magee DJ, 2008). In 1947, Adson first described this test with the explanation that an alteration of the radial pulse or an alteration in blood pressure is considered a pathognomonic sign of scalenus anticus syndrome indicating that the vascular component of neurovascular bundle is compressed by scalenus anticus muscle. (Mackinnon SE, 2002)

Halstead Maneuver (See picture appendix 4): The Reverse-Adson Maneuver, or Halstead Maneuver, is also done with the patient's arm externally rotated and extended with the elbow extended. The examiner monitors the radial pulse as the patient rotates the head away from the affected side and extends the neck. The patient is instructed to take a deep breath and hold it. The absence or disappearance of a pulse indicates a positive test a suggesting the presence of a cervical rib (Magee DJ, 2008)

Roos Test (See picture appendix 5): This test will be used to screen interested participants during the recruitment phase. The patient stands and abducts the arms to 90 degrees, externally rotates the shoulder and flexes the elbows to 90 degrees. The patient is then directed to open and close the hands slowly for three minutes. A positive test will cause increased symptoms such as ischemic pain, heaviness or profound weakness of the arm or numbness and tingling of the hand. Minor fatigue is considered a negative test. (Magee DJ, 2008) Positive findings indicate compression of the neurovascular bundle specific to structures in the thoracic outlet.

In previous studies testing the efficacy of the TOS special tests, Doppler ultrasonography was shown to visualize vascular abnormalities and confirmed the diagnosis in patients with at least five positive provocative (special) tests. (Gillard, Perez-Cousin, Hachulla, Remy et al 2001). Our research team would like to confirm this previous finding and further expand on this topic by examining for the changes in blood flow with Doppler ultrasonography during the performance of these special tests.

Diagnostic ultrasound has been in use since the late 1950s. There are no confirmed adverse biological effects on patients from this usage. Although no hazard has been identified that would limit the use of diagnostic ultrasound on patients in education and research, experience from normal diagnostic practice may or may not experience hazards due to extended exposure times and altered conditions. Participants enrolled in this study will be informed about the anticipated exposure conditions and how these compare with normal diagnostic practice (AIUM, 2007).

In addition to evaluation of the effectiveness of the TOS special tests, the effects of Osteopathic manipulative treatment (OMT) to help alleviate TOS symptoms is also of interest. OMT of TOS is directed towards improving mechanics of the cervical, upper thoracic spine, upper ribs, clavicles and muscles of the neck, shoulder and pectoral girdle. OMT procedures such as myofascial release and articulatory techniques can be useful in reducing the dysfunctions of these regions which is causing compression on the nerve. Myofascial release involves manipulating the soft tissues, articulation is taking a joint through its available range of motion to improve its normal physiological movement (Ward, 2003). By performing this research we can improve the body of research in osteopathic manipulative medicine (OMM) and provide a proven means of treating the pain experienced by individuals with TOS.

TOS diagnosis and treatment is taught to osteopathic medical students, physical therapy students as well as other health professionals that employ manual therapy strategies to diagnose and treat musculoskeletal disorders. Despite this information being included as part of the education of these health care professionals, there is little literature outside of patient anecdotes that supports the reliability and validity of these tests and treatments. We hope to contribute towards increasing the evidence of these tests and treatments for TOS to ensure that students especially those at the health professions division at NSU will be educated on reliable and proven orthopaedic/special tests and to extrapolate our results to all educators and health care professionals that diagnose TOS.

In today's hectic society it becomes a great disadvantage to individuals when they develop pain and discomfort that decreases their ability to function efficiently. Thoracic Outlet Syndrome (TOS) is a condition that causes pain in the upper extremity, typically extending along the inner aspect of the arm and hand. Other symptoms include weakness, numbness and tingling in the upper extremity. A neurovascular bundle that consists of the brachial plexus, subclavian artery and vein travels from the neck into the arm. TOS symptoms result when the nerves or blood vessels are compressed by the surrounding anatomical structures. In performing this research study, our team would like to improve awareness of TOS to all health care professionals as an entrapment neuropathy and differential diagnosis to neck pain with referred pain. We would also like to bring osteopathic medicine, physical therapy and other paradigms of musculoskeletal manual medicine/therapy together to develop a standardized and valid approach to the diagnosis and treatment of TOS which is not currently available.

There are multiple possible causes of TOS, majority of which results in anatomic restrictions. These possible causes include trauma to the shoulder girdle and more commonly postural disturbances. Individuals with TOS often sit at a computer or desk for an extended period of time for work or school. They develop rounded shoulders and a forward head carriage which changes the length and tone of certain muscles and the relationship of structures in relation to the neurovascular bundle. The anatomic disturbances that contribute and is of the greatest interest to osteopathy includes hypertonicity of the anterior and middle scalene muscles in the neck, hypertonicity of the pectorialis muscle from the upper extremity to the 3-5th ribs, somatic dysfunctions of the clavicle, upper thoracic region and ribs (especially the first rib) (Ward, 2003).

TOS is often the resulting diagnosis after elimination of other possible conditions that cause similar symptoms. These other possible conditions include disc herniations, osteoarthritis, tumors and nerve entrapment syndromes such as carpal tunnel syndrome. Currently discrepancies exist between clinicians about the correct approaches to diagnosis and treatment of TOS. Today's technological advancements can help provide more information about the patient's anatomy, however none can be used for diagnosis alone. MRIs are usually best used for confirmation for the evaluation of the region of interest, however in TOS, findings are frequently inconclusive. One reason for this may be the difficulty to evaluate the extent of a muscle spasm or rib somatic dysfunction and the degree to which it is compressing a nerve structure. (Koknel 2005). X-rays are used to eliminate extra ribs in the cervical region as a cause for symptoms. Anomalous cervical ribs are found in 0.17% to 0.74% each year, however, only 10% of individuals experience TOS symptoms and the onset of these symptoms often relates to cervical spine trauma (Novak, Mackinnon, 2002). The diagnosis of TOS remains to be best based on the patient's subjective complaints, physical examination and the exclusion of other pathologies (Novak, Mackinnon, 2002). Clinical assessment of TOS is best achieved by reproduction of symptoms with compression and special orthopaedic provocative tests that re-produces symptoms based on patient position (Koknel, 2005).

These orthopedic special tests will include:

Wright Test: Wright Test, or Hyperabduction Test, is done by bringing the arm into full abduction with the shoulder externally rotated and the elbow extended while monitoring the radial pulse throughout (Magee DJ, 2008). If there is a decrease or absence of pulse the test is positive showing that axillary artery is compressed by either the pectoralis minor muscle or the coracoid process. (Köknel Talu G, 2005)

Adson Test: For Adson Maneuver the examiner externally rotates and extends the effected arm with the elbow extended while monitoring the radial pulse. The patient is then instructed to rotate the head toward the affected side, extend the neck and take a deep breath and hold it. The absence of disappearance of a pulse indicates a positive test (Magee DJ, 2008). In 1947, Adson first described this test with the explanation that an alteration of the radial pulse or an alteration in blood pressure is considered a pathognomonic sign of scalenus anticus syndrome indicating that the vascular component of neurovascular bundle is compressed by scalenus anticus muscle. (Mackinnon SE, 2002)

Halstead Maneuver: The Reverse-Adson Maneuver, or Halstead Maneuver, is also done with the patient's arm externally rotated and extended with the elbow extended. The examiner monitors the radial pulse as the patient rotates the head away from the affected side and extends the neck. The patient is instructed to take a deep breath and hold it. The absence or disappearance of a pulse indicates a positive test a suggesting the presence of a cervical rib (Magee DJ, 2008)

Roos Test: This test will be used to screen interested participants during the recruitment phase. The patient stands and abducts the arms to 90 degrees, externally rotates the shoulder and flexes the elbows to 90 degrees. The patient is then directed to open and close the hands slowly for three minutes. A positive test will cause increased symptoms such as ischemic pain, heaviness or profound weakness of the arm or numbness and tingling of the hand. Minor fatigue is considered a negative test. (Magee DJ, 2008) Positive findings indicate compression of the neurovascular bundle specific to structures in the thoracic outlet.

In previous studies testing the efficacy of the TOS special tests, Doppler ultrasonography was shown to visualize vascular abnormalities and confirmed the diagnosis in patients with at least five positive provocative (special) tests. (Gillard, Perez-Cousin, Hachulla, Remy et al 2001). Our research team would like to confirm this previous finding and further expand on this topic by examining for the changes in blood flow with Doppler ultrasonography during the performance of these special tests.

Diagnostic ultrasound has been in use since the late 1950s. There are no confirmed adverse biological effects on patients from this usage. Although no hazard has been identified that would limit the use of diagnostic ultrasound on patients in education and research, experience from normal diagnostic practice may or may not experience hazards due to extended exposure times and altered conditions. Participants enrolled in this study will be informed about the anticipated exposure conditions and how these compare with normal diagnostic practice (AIUM, 2007).

In addition to evaluation of the effectiveness of the TOS special tests, the effects of Osteopathic manipulative treatment (OMT) to help alleviate TOS symptoms is also of interest. OMT of TOS is directed towards improving mechanics of the cervical, upper thoracic spine, upper ribs, clavicles and muscles of the neck, shoulder and pectoral girdle. OMT procedures such as myofascial release and articulatory techniques can be useful in reducing the dysfunctions of these regions which is causing compression on the nerve. Myofascial release involves manipulating the soft tissues, articulation is taking a joint through its available range of motion to improve its normal physiological movement (Ward, 2003). By performing this research we can improve the body of research in osteopathic manipulative medicine (OMM) and provide a proven means of treating the pain experienced by individuals with TOS.

TOS diagnosis and treatment is taught to osteopathic medical students, physical therapy students as well as other health professionals that employ manual therapy strategies to diagnose and treat musculoskeletal disorders. Despite this information being included as part of the education of these health care professionals, there is little literature outside of patient anecdotes that supports the reliability and validity of these tests and treatments. We hope to contribute towards increasing the evidence of these tests and treatments for TOS to ensure that students especially those at the health professions division at NSU will be educated on reliable and proven orthopaedic/special tests and to extrapolate our results to all educators and health care professionals that diagnose TOS.

ELIGIBILITY:
Inclusion Criteria:

* positive Roo's test indicative of thoracic outlet syndrome
* one positive provocative test for thoracic outlet syndrome from:Adson's, Wright's or Halstead's indicative of the specific tissue that is impeding blood flow to the upper extremity.

Exclusion Criteria:

* known medical history of cervical disc disease (such as herniated discs, degenerative disc disease
* known medical history of upper extremity nerve entrapment syndromes such as carpal tunnel syndrome, pronator teres syndrome, anterior interosseus syndrome, ulnar groove, cubital tunnel, Guyon's canal or radial tunnel syndrome.
* medical history of diabetic/thyroid related neuropathies and medicine induced paresthesias
* medical history of atherosclerosis or any type of clotting or other vascular disorders such as thromboembolism of the upper extremity
* excessive pain during Patients with excessive pain during passive shoulder range of motion procedures such as in 'frozen shoulder'

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from a variety of settings:
  1. First and second year medical students from Nova Southeastern University College of Osteopathic Medicine with symptoms of Thoracic outlet syndrome.
  2. Patients from the Sanford Ziff Osteopathic Manipulation Clinic that exhibit symptoms of Thoracic outlet syndrome
  3. Patients from the Nova Southeastern University Sports Medicine Clinic that exhibit symptoms of Thoracic outlest syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood flow velocity | 5 minutes
  Doppler ultrasound was utilized to measure blood flow velocity during TOS special tests pre and post osteopathic manipulative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Qureshi, DPT, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States